CLINICAL TRIAL: NCT06497153
Title: Lung Ultrasound in Pediatric Acute Chest Syndrome
Acronym: Lupacs
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240137; IDRCB: 2023-A02741-44 (Other: ANSM)
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Sickle Cell Disease
Keywords: acute chest syndrome; lung ultrasound; LUS score; ventilation; clinical severity
MeSH Terms: conditions — Anemia, Sickle Cell; Acute Chest Syndrome; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sickle cell anaemia patients with acute chest syndrome
  Interventions: Procedure: lung ultrasound

INTERVENTIONS:
Procedure: lung ultrasound — lung ultrasound repeated according to protocol during the stay in the paediatric intensive care unit

SUMMARY:
Sickle-cell disease is a common disease with serious complications, in particular acute chest syndrome (ACS), which can be life threatening. The pathophysiology of ACS is poorly understood, but alveolar hypoventilation appears to play an important role. Pulmonary ultrasound is increasingly used in pediatrics to diagnose ACS. The management of ACS is complex, including oxygen therapy, antibiotics, spirometry, transfusions and ventilatory support. ACS and acute vaso-occlusive pain are the main reasons for hospitalisation in pediatric intensive care units. The aim of this study was to identify the pulmonary indicators correlated with ventilation time in these children, and to study the correlations between the results of lung ultrasound (LUS) and the clinical severity of the episode. The inclusion criteria for this study are the presence of an ACS in a child aged between 1 month and 17 years hospitalised in the pediatric intensive care unit at Robert-Debre Hospital who has not expressed any opposition and without opposition from their legal representative. The study will run for 2 years, with a target of 60 patients. Each patient included in the study will have multiple LUS during their care, in accordance with a protocol, and their clinical, biological and radiological data will be collected during their stay in the department.

DETAILED DESCRIPTION:
Scientific rationale: Sickle-cell disease is a frequent disorder with a high morbidity. Its course is marked by acute complications with a life-threatening and functional prognosis, principally acute chest syndrome (ACS). This syndrome is caused by a combination of infection, fat embolism, and vaso-occlusion of the pulmonary vasculature. The pathophysiology of this syndrome is poorly understood, although alveolar hypoventilation plays an important role in its genesis. Pulmonary ultrasound is being used exponentially in pediatrics, and several studies have shown that it performs well in diagnosing ACS. Bedside lung ultrasound scans are now routinely performed in the management of patients with suspected or confirmed ACS. The management of ACS is multimodal, with the use of oxygen, antibiotics, incentive spirometry, transfusions, exchange transfusions and ventilatory assistance. Along with acute vaso-occlusive pain, ACS in children with sickle cell disease is the main reason for admission in pediatric intensive care. There are no recommendations concerning ventilatory support or transfusion in this situation. Lung parenchymal aeration and its evolution, as assessed by lung ultrasound, may allow patients to be categorised and ventilatory strategies and transfusion adapted.

Objective and primary endpoint:

- To identify the indicator of lung involvement assessed by LUS that best correlates with ventilation time in children with sickle cell disease admitted to the pediatric intensive care unit with suspected ACS.

Objectives and secondary endpoints:

* To study the correlation between LUS score and other markers of the clinical severity of the episode (invasive and non-invasive ventilation parameters, maximal FiO2, maximal PCO2, transfusion).
* To study the correlation between LUS score and clinical score (correlation with the Clinical Respiratory Score (CRS) and pulmonary auscultation).

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease patient aged 1 month to 17 years
* Hospitalisation in the PICU of Robert-Debre hospital
* Suspicion of acute chest syndrome ACS
* No objection from a legal representative or the child taken in by the doctor.

Exclusion Criteria:

* Refusal of parents
* Delay between first LUS and initiation of ventilator support greater than 6 hours
* Patient without social insurance

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Acute Chest Syndrome in sickle cell patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficients between LUS scores (lung ultrasound) at H0, H8, H24, H48, H72 and duration of ventilation (invasive and non-invasive combined) | length of stay in intensive care unit (15 days)

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie HAYOTTE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré hOSPITAL, Paris, France